CLINICAL TRIAL: NCT04176796
Title: Don't Throw Your Heart Away: Medical Student Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Gretchen Chapman, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1 F30 HL152526-01-B; 20PRE35120492 (Other Grant/Funding Number: American Heart Association); 1F30HL152526-01 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Transplant Disorder
Keywords: Heart Transplant; Transplant Survival; Applied Ethics; Medical Students; Human Behavior; Decision Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1: Combined only (No Intervention): Participants randomized to baseline (control) arm Condition 1 will view only combined transplant survival outcome information (e.g. transplant survival rate not stratified by number and quality of donor hearts accepted at each center) when making a choice between the two hospitals.
- Condition 3: Stratified only (Experimental): Participants randomized to Condition 3 will view only stratified transplant survival outcome information when making a choice between the two hospitals.
  Interventions: Other: Stratified Transplant Survival

INTERVENTIONS:
Other: Stratified Transplant Survival — The transplant survival rate in the table of outcome statistics is stratified into two groups: (i) patients who received excellent donor organs and (ii) patients who received less than optimal donor organs.
  Stratified transplant survival is computed from survival rates of transplant patients who received each quality category of organ.
  excellent transplant survival = [number of patients surviving after transplant with excellent organ]/[number of patients for whom excellent organ was accepted for transplant] marginal transplant survival = [number of patients surviving after transplant with marginal organ]/[number of patients for whom marginal organ was accepted for transplant]
  Arms: Condition 3: Stratified only

SUMMARY:
Publicly available outcome assessments for transplant programs do not make salient that some programs tend to reject many of the hearts they are offered, whereas other programs accept a broader range of donor offers. The investigators use empirical studies to test whether transplant center performance data (i.e. transplant and waitlist outcome statistics) that reflect center donor acceptance rates influence laypersons to evaluate centers with high organ decline rates less favorably than centers with low organ decline rates. 125 medical student participants will be recruited from University of Pittsburgh Medical School and randomized to one of two different information presentation conditions. Participants will be given an introduction to the donor organ match process, then asked to view the table of transplant outcomes corresponding to the condition they were randomized to. Each participant is asked to choose the hospital that they would consider to be "higher performing" between two hospitals: one hospital with a non-selective, "accepting" strategy (takes all donor heart offers), and one hospital with a more selective, "cherrypicking" strategy (tends to reject donor offers that are less than "excellent" quality).

DETAILED DESCRIPTION:
Publicly available outcome assessments for transplant programs do not make salient that some programs tend to reject many of the hearts they are offered, whereas other programs accept a broader range of donor offers. The investigators use empirical studies to test whether transplant center performance data (i.e. transplant and waitlist outcome statistics) that reflect center donor acceptance rates influence laypersons to evaluate centers with high organ decline rates less favorably than centers with low organ decline rates. 125 medical student participants will be recruited from University of Pittsburgh Medical School and randomized to one of two different information presentation conditions:

Condition 1 ("baseline" condition): view only combined transplant survival (e.g. transplant survival rate not stratified by number and quality of donor hearts accepted at each center)

Condition 2: view only stratified transplant survival (e.g. transplant survival rate stratified into patients who received excellent donor organs and patients who received less than optimal donor organs)

Participants will be given an introduction to the donor organ match process, then asked to view the table of transplant outcomes corresponding to the condition they were randomized to.Each participant is asked to choose the hospital that they would consider to be "higher performing" between two hospitals: one hospital with a non-selective, "accepting" strategy (takes all donor heart offers), and one hospital with a more selective, "cherrypicking" strategy (tends to reject donor offers that are less than "excellent" quality). In order to identify the decision process that underlies this choice pattern, the investigators will examine a putative mediator. Specifically, participants will be asked to rate the extent to which they considered patients' chances of getting an excellent heart, avoiding a less-than-optimal heart, and getting any type of heart when making their choice between the two hospitals.

ELIGIBILITY:
Inclusion Criteria:

Participants will be asked to participate if they confirm the following inclusion criteria in the consent form.

1. 18 years of age or older
2. must read and understand the information in the consent form
3. must want to participate in the research and continue with the survey
4. must live in United States
5. 2nd, 3rd, or 4th year medical student at University of Pittsburgh School of Medicine

Exclusion Criteria:

1. participants who do not meet primary criterion of being a 2nd, 3rd, or 4th year medical student at University of Pittsburgh School of Medicine

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Butler, BS, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will make all of the raw IPD files - together with statistical analysis protocol descriptions and information for proper analysis available for download a minimum of 1 year, and a maximum of 3 years, after publication of the corresponding manuscripts. All human subjects data are anonymized immediately when they are initially written from the online survey platform to the server, and thus participant confidentiality will not be compromised by this plan for data sharing.
  All hypotheses, methods, and planned analyses for the applicant's studies will be pre-registered on ClinicalTrials.gov and Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All of the raw files, statistical analysis protocol descriptions, and information for proper analysis will be available for download a minimum of 1 year, and a maximum of 3 years, after publication of the corresponding manuscripts.
URL: https://osf.io/9fsb3/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited via email through medical school listserv.
Pre-assignment Details: Included if the participant identified as current medical student and was over 18.
Groups:
- Condition 3: Stratified Only: Participants randomized to Condition 3 will view only stratified transplant survival outcome information when making a choice between the two hospitals.
  Stratified Transplant Survival: The transplant survival rate in the table of outcome statistics is stratified into two groups: (i) patients who received excellent donor organs and (ii) patients who received less than optimal donor organs.
  Stratified transplant survival is computed from survival rates of transplant patients who received each quality category of organ.
  excellent transplant survival = [number of patients surviving after transplant with excellent organ]/[number of patients for whom excellent organ was accepted for transplant] marginal transplant survival = [number of patients surviving after transplant with marginal organ]/[number of patients for whom marginal organ was accepted for transplant]
Period: Overall Study
Arm/Group | Condition 1: Combined Only | Condition 3: Stratified Only
Started | 56 | 49
Completed | 56 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Medical trainees
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1: Combined Only | Condition 3: Stratified Only | Total
Number analyzed (Participants) | 56 | 49 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 49 | 105
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 37 | 30 | 67
  Male | 19 | 17 | 36
  Transgender | 0 | 1 | 1
  Unknown | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 8 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 33 | 36 | 69
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 56 | 49 | 105

OUTCOME MEASURES:

1. Primary Outcome: Hospital Choice
Description: The outcome variable will be a measure of binary choice between two hospitals: one with a selective donor-heart acceptance strategy and one with a non-selective donor heart acceptance strategy.
  Participants will respond to the question "Which Hospital is a better choice for patients? Please click on one of the two tables below to indicate which hospital is the better choice." Participants will choose been two outcome tables featuring the selective and non-selective hospital (counterbalanced, such that each of the two choices is equally likely to be presented at top of the choice scenario in each condition). The number of participants that choose each hospital will be the measured outcome variable used in analyses.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Condition 1: Combined Only | Condition 3: Stratified Only
Number analyzed (Participants) | 56 | 49
Participants
  Number choosing non-selective center | 33 | 47
  Number choosing selective center | 23 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Condition 1: Combined Only | Condition 3: Stratified Only
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/49
Other Adverse Events (participants affected / at risk) | 0/56 | 0/49

LIMITATIONS AND CAVEATS:
Selection bias from use of medical school listserv to recruit trainees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04176796/Prot_SAP_000.pdf